CLINICAL TRIAL: NCT00646308
Title: Assessment of Cardiovascular Risk Markers in GH Deficient Patients With Nonsecreting Pituitary Adenomas
Brief Title: Assessment of Cardiovascular Risk Markers in Growth Hormone Deficient Patients With Nonsecreting Pituitary Adenomas
Status: Terminated | Type: Observational
Why Stopped: Poor enrollment
Sponsor: Columbia University (Other)
Collaborators: EMD Serono (Industry); Genentech, Inc. (Industry)
Responsible Party: Pamela U. Freda MD, Columbia Univesrity
Other Study IDs: AAAB9681
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Growth Hormone Deficiency; Pituitary Tumor
Keywords: growth hormone deficiency, pituitary tumors
MeSH Terms: conditions — Dwarfism, Pituitary; Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- I: Adult patients with GH deficiency due to a nonsecreting pituitary tumor
- 2: Adult patients with a nonsecreting pituitary tumor but without GH deficiency

SUMMARY:
The purpose of this study is to determine if patients with a history of nonsecreting pituitary adenomas with untreated GH deﬁcient patients have proﬁles consistent with increased cardiovascular risk compared to patients without GH deficiency who have undergone similar surgery.

DETAILED DESCRIPTION:
PROJECT TITLE: Assessment of Cardiovascular Risk in Patients with Growth Hormone Deficiency Following Transsphenoidal Surgery for Nonsecreting Pituitary Adenomas.

BACKGROUND Recently, an awareness of the risks of hypopituitarism in adults has been raised by epidemiological studies demonstrating its association with increased mortality, likely from cardiovascular (CV) causes. In particular, untreated growth hormone deficiency has been implicated as a possible cause of this increased mortality. A 2004 clinical review of growth hormone deficiency in adults highlights the plausibility of this argument by citing studies potentially linking GHD to the following: elevated CRP, LDL and coagulation factor levels, increased abdominal obesity, increased insulin resistance, increased prevalence of structural and functional heart disease and increased rates of endothelial cell and large artery dysfunction. Furthermore, therapy for GH deficiency has been shown to lower total and LDL cholesterol and reduce visceral fat mass, reduce signs of early atherosclerosis and perhaps decrease overall risk of myocardial infarction. While these studies suggest that GHD is an important cardiovascular risk factor, we believe the data are imperfect since some of the studies chose comparison groups too dissimilar (allowing for the possibility of unrecognized confounding). Previous studies have assessed cardiovascular risk in patients with hypopituitarism in comparison to the general population or much younger GH replaced subjects or GHD patients before and after GH therapy. In contrast, we plan to compare cardiovascular risk among adult patients rendered growth hormone deficient following surgery for a non secreting pituitary adenoma versus patients who have undergone the same surgery but who remain growth hormone sufficient. We plan to test for growth hormone deficiency using the Arginine/GHRH stimulation test in 80 subjects. We will divide the patients into two groups: growth hormone deficient and growth hormone sufficient. Once we have recruited enough patients in each group (thirty), we will compare known CV risk markers and endothelial function in carefully matched patients from each group. This approach will allow us to compare similar patients (i.e. all will have undergone surgery, some in each group will have undergone radiation) whose primary difference will be the GH status. In addition, from each group we will identify patients with additional pituitary deficiencies in the hope of comparing patients with either isolated GHD or patients with multiple endocrinopathies to similar matched controls.

At least two other novel aspects of our study include the use of magnetic resonance spectroscopy to measure intramyocellular and intrahepatic lipids and venous endothelial cell biopsy to assess endothelial function. Regarding the first modality, elevated levels of intramyocellular and intrahepatic lipids have been associated with insulin resistance in other populations. It is our hypothesis that subtle abnormalities in these lipid stores may correlate with insulin resistance in patients with apparent occult GH deficiency. With regard to endothelial function, previous work has linked GHD with endothelial cell dysfunction but typically through indirect measures including serum markers and arterial flow mediated dilatation. However, a technique has been recently developed to safely sample venous endothelial cells which in turn will enable us to assess directly at the level of endothelial cells, oxidative stress, cell activation and nitric oxide synthesis. It is our belief that this new method will help confirm the contention that GHD alters the basic function of endothelial cells.

STUDY DESIGN This study will assess the level of cardiovascular risk in two patient populations: those patients who are GHD following transsphenoidal surgery for nonsecreting pituitary adenomas and those patients who are not GHD following similar surgery. The primary outcome will be serum markers of cardiovascular risk including lipids, CRP, IL6 and homocysteine.

Experimental Protocol:

Subjects for this study will have all undergone transsphenoidal surgery for a nonsecreting pituitary adenoma. In addition, there may be some additional subjects, who have also undergone transsphenoidal surgery for a nonsecreting pituitary adenoma, recruited by word of mouth from the cohort of patients described above. Only patients who are not receiving GH therapy will be considered. Of those patients who have received RT, only those at least 5 years from radiotherapy will be recruited in order to lessen the likelihood of a false positive Arginine/GHRH stimulation test which can occur in the early years post RT.

The remaining respondents will be stratified into two groups based on the presence or absence of a history of other hypopituitarism: 1) those with > 1 known pituitary hormone deficiency (other than GH) and who are on replacement for these and 2) those with no known pituitary hormone deficits. The status of other pituitary hormone replacement therapies will be verified prior to the arrival of the subjects for further testing. Patients will need to be on stable doses of replacement therapy for at least 3 months prior to the study visit and if on hormone replacements they must be on hydrocortisone < 30 mg/day or equivalent and physiological doses of thyroid and sex steroid replacements. If possible, patients will be asked to provide copies of their most recent endocrine studies if these were not available from the chart review to verify the adequacy of their replacement therapy. Any woman known to be pregnant or any woman of childbearing age with a positive urinary HCG will not be considered for the study (we will screen all woman of childbearing age at the first visit prior to initiation of any testing). In addition, any woman actively nursing cannot be included in the study (we will ask all women of childbearing age at the first visit). We will recruit equal numbers from these two groups, inviting subjects to our Neuroendocrine Unit for an initial visit where they will undergo a clinical exam with vital signs, anthropometric measurements and skin fold thickness assessments. Subjects will also undergo GH stimulation testing with Arginine/GHRH to identify GH deficient (peak GH < 4 µg/L) and nonGH de•cient (peak GH > 10 µg/L) groups. Lastly, all subjects will have an endothelial cell biopsy performed.

Thirty matched pairs of patients from the GHD and GH sufficient groups will be contacted further for an additional visit to our unit for some or all of the following tests:

* Fasting blood sampling for CV risk markers including CRP, homocysteine, lipoproteins, IL6 IGFI and IGFBP3 (all subjects, n=30 pairs)
* 75 gm OGTT; Insulin and glucose (all subjects, n=30 pairs)
* DEXA scan to assess body composition and bone density (all subjects, n=30 pairs)
* Ultrasound to assess carotid intimal medial thickness and brachial artery flowmediated dilatation (subset of subjects, n=10 pairs).
* Magnetic resonance spectroscopy assessment of intramyocellular lipids and intrahepatic lipids in a subset of each group of the cohort (subset of subjects, n=10 pairs). Subjects will be studied within 6 months of their initial GH stimulation test.

STUDY DRUGS Subjects will undergo an Arginine/GHRH stimulation test. They will receive Rgene (Upjohn) a 10% Arginine Hydrochloride solution in water and Geref Diagnostic (Serono).

STUDY SUBJECTS Subjects for the study will include adult patients who have undergone transsphenoidal pituitary surgery for a nonsecreting pituitary adenoma.

STUDY LOCATION This study will take place out of the Neuroendocrine Unit, Columbia University.

POTENTIAL RISKS Participation in this study will involve minimal standard risks associated with blood draws. In addition there is a potential risk from exposure to radiation from DEXA scans. However, the amount of radiation exposure from DEXA scanning is only one percent of a chest xray and it is in accordance with federal guidelines for this type of research. Given the risk posed to a fetus from radiation exposure, pregnant or nursing mothers will be excluded from the study. To assess for pregnancy we will chec a urine HCG on all women of childbearing age prior to initiating any testing. In addition, women of childbearing age will be asked if they actively nursing and if so they will be excluded from the study. Since the risk to pregnant or nursing mothers is present only at the time of testing, no additional precautions against pregnancy need to be taken in the days following our testing. Ultrasound (for IMT and flow mediated dilatation studies) poses minimal risk beyond mild discomfort from the gel and probe. MRI also poses minimal risk beyond mild discomfort from the enclosed space and noise of the machine as long as there is no metal within the scanner room. The subjects will be asked a series of questions by the MRI technicians to ensure that they are safe to proceed with MRI. In addition, pregnant woman cannot undergo MRI. The risks of endothelial biopsy are thought to include pain, inflammation, infection and clots. In a previous study it was found to be safe but patients will be asked to return one week after the biopsy for evaluation of the site. If any symptoms arise prior to one week follow up patients will be advised to call or proceed to the emergency room.

The most common adverse reactions from the administration of arginine include nausea, vomiting, headache, flushing, numbness, local venous irritation. Systemic allergic reaction is rare but patients with highly allergic tendencies will not be included. Pregnant or nursing subjects will also be excluded as mentioned above. For GHRH, common side effects include transient warmth/flushing of face, injection site pain, redness/swelling at site of injection, nausea, headache, vomiting, strange taste in mouth, paleness, tightness in chest. A physician will be present throughout the administration of these two drugs.

POTENTIAL BENEFITS The results of the growth hormone stimulation test will be made available to subjects and their doctors. Therefore, if a subject is found to be growth hormone deficient, he or she might benefit from growth hormone therapy which has been shown, in some studies, to improve body composition, cholesterol levels and other factors associated with an increased risk for cardiovascular disease. A decision to initiate therapy, however should only occur after a careful discussion between the subject and his or her personal physician occurs. There may also be some benefit from DEXA scanning as it might identify previously undiagnosed osteoporosis. This condition has effective treatment options. Lastly, participation in the study will help further contribute to our understanding of the risk of heart disease in growth hormone deficient patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a history of a nonsecreting pituitary tumor with or without prior pituitary surgery.

Exclusion Criteria:

* Current use of GH therapy or within the prior 3 months. Pituitary tumor necessitating surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a history of nonsecreting pituitary tumor.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Cardiovascular risk markers, speciﬁcally lipids, CRP, IL6 and homocysteine | One time point

SECONDARY OUTCOMES:
Total body fat, trunk fat and lean body mass by DEXA, insulin sensitivity, flow mediated dilatation and endothelial cell biopsy, carotid IMT, intramyocellular and intrahepatic lipid content. | One time point

CONTACTS AND LOCATIONS:
Overall Officials: Pamela U Freda, MD, Principal Investigator — Columbia University College of P & S
Locations (1):
- Columbia University Neuroendocrine Unit, New York, New York, United States